CLINICAL TRIAL: NCT01696266
Title: An International Survey on Hypoglycaemia Among Insulin-treated Patients With Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-4019; U1111-1132-1910 (Other: WHO)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin-treated patients with diabetes
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Patients will be asked to complete a two-part patient self-assessment questionnaire (SAQ) comprising a retrospective cross-sectional evaluation (Part 1), and a prospective observational evaluation (Part 2).

SUMMARY:
This study is conducted in Europe. The aim of the study is to gather information about hypoglycaemia (low blood glucose) among patients with Type 1 or Type 2 diabetes mellitus. The study is both retrospective and prospective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 diabetes mellitus treated with insulin for more than 12 months
* Patients giving informed consent to participate in the survey

Exclusion Criteria:

* Non-ambulatory patients
* Illiterate patients and patients otherwise unable to complete a written survey

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Insulin-treated patients with Type 1 or Type 2 diabetes mellitus. Patients should be ambulatory, literate, have used insulin for at least 12 months, and be over 18 years of age to be able to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 29304 (Actual)
Dates: Start 2012-09-05 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2013-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of any hypoglycaemic event | In the 4 weeks prior to and following the baseline visit (Week 0)

SECONDARY OUTCOMES:
Difference in the reported incidence rates of any hypoglycaemia | In the 4 weeks prior to (Part 1) versus following (Part 2) the baseline visit
Incidence of hypoglycaemic events requiring hospital admission | In the 6 months prior to and 4 weeks following the baseline visit
Incidence of all severe hypoglycaemic events | In the 6 months prior to and 4 weeks following the baseline visit
Incidence of probable symptomatic hypoglycaemic events | In the 4 weeks prior to and following the baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (24):
- Novo Nordisk Investigational Site, Prov. de Buenos Aires, Argentina
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Novo Nordisk Investigational Site, Prague, Czechia
- Novo Nordisk Investigational Site, Copenhagen S, Denmark
- Novo Nordisk Investigational Site, Espoo, Finland
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Budapest, Hungary
- Novo Nordisk Investigational Site, Bangalore, India
- Novo Nordisk Investigational Site, Kfar Saba, Israel
- Novo Nordisk Investigational Site, Amman, Lebanon
- Novo Nordisk Investigational Site, Selangor Darul Ehsan, Malaysia
- Novo Nordisk Investigational Site, Mexico City, Mexico
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands
- Novo Nordisk Investigational Site, Warsaw, Poland
- Novo Nordisk Investigational Site, Bucharest, Romania
- Novo Nordisk Investigational Site, Moscow, Russia
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Belgrade, Serbia
- Novo Nordisk Investigational Site, Bratislava, Slovakia
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- Novo Nordisk Investigational Site, Malmo, Sweden

REFERENCES:
- [Result] Khunti K, Alsifri S, Aronson R, Cigrovski Berkovic M, Enters-Weijnen C, Forsen T, Galstyan G, Geelhoed-Duijvestijn P, Goldfracht M, Gydesen H, Kapur R, Lalic N, Ludvik B, Moberg E, Pedersen-Bjergaard U, Ramachandran A; HAT Investigator Group. Rates and predictors of hypoglycaemia in 27 585 people from 24 countries with insulin-treated type 1 and type 2 diabetes: the global HAT study. Diabetes Obes Metab. 2016 Sep;18(9):907-15. doi: 10.1111/dom.12689. Epub 2016 Jun 20. PMID 27161418
- [Result] Khunti K, Alsifri S, Aronson R, Cigrovski Berkovic M, Enters-Weijnen C, Forsen T, Galstyan G, Geelhoed-Duijvestijn P, Goldfracht M, Gydesen H, Kapur R, Lalic N, Ludvik B, Moberg E, Pedersen-Bjergaard U, Ramachandran A; HAT Investigator Group. Impact of hypoglycaemia on patient-reported outcomes from a global, 24-country study of 27,585 people with type 1 and insulin-treated type 2 diabetes. Diabetes Res Clin Pract. 2017 Aug;130:121-129. doi: 10.1016/j.diabres.2017.05.004. Epub 2017 May 12. PMID 28602812
- [Result] Kern W, Holstein A, Moenninghoff C, Kienhofer J, Riedl M, Kulzer B. Self-reported Hypoglycaemic Events in 2 430 Patients with Insulin-treated Diabetes in the German Sub-population of the HAT Study. Exp Clin Endocrinol Diabetes. 2017 Oct;125(9):592-597. doi: 10.1055/s-0043-112350. Epub 2017 Jul 27. PMID 28750429
- [Result] Pongrac Barlovic D, Zavratnik A, Skvarca A, Jansa K, Vukelic B, Tomazic M, Ravnik Oblak M. Self-reported Hypoglycaemia in Patients treated with Insulin: A Large Slovenian Retrospectively-prospective Study. Zdr Varst. 2017 Oct 9;56(4):244-250. doi: 10.1515/sjph-2017-0033. eCollection 2017 Oct. PMID 29062399
- [Result] Aronson R, Goldenberg R, Boras D, Skovgaard R, Bajaj H. The Canadian Hypoglycemia Assessment Tool Program: Insights Into Rates and Implications of Hypoglycemia From an Observational Study. Can J Diabetes. 2018 Feb;42(1):11-17. doi: 10.1016/j.jcjd.2017.01.007. Epub 2017 May 17. PMID 28528246
- [Result] Hussein Z, Kamaruddin NA, Chan SP, Jain A, Uppal S, Bebakar WMW; HAT study investigators in Malaysia. Hypoglycemia awareness among insulin-treated patients with diabetes in Malaysia: A cohort subanalysis of the HAT study. Diabetes Res Clin Pract. 2017 Nov;133:40-49. doi: 10.1016/j.diabres.2017.08.007. Epub 2017 Aug 14. PMID 28888148
- [Result] Aronson R, Galstyan G, Goldfracht M, Al Sifri S, Elliott L, Khunti K. Direct and indirect health economic impact of hypoglycaemia in a global population of patients with insulin-treated diabetes. Diabetes Res Clin Pract. 2018 Apr;138:35-43. doi: 10.1016/j.diabres.2018.01.007. Epub 2018 Jan 31. PMID 29355651
- [Result] Haluzik M, Kretowski A, Strojek K, Czupryniak L, Janez A, Kempler P, Andel M, Tankova T, Boyanov M, Smircic Duvnjak L, Madacsy L, Tarnowska I, Zychma M, Lalic N. Perspectives of Patients with Insulin-Treated Type 1 and Type 2 Diabetes on Hypoglycemia: Results of the HAT Observational Study in Central and Eastern European Countries. Diabetes Ther. 2018 Apr;9(2):727-741. doi: 10.1007/s13300-018-0388-2. Epub 2018 Mar 9. PMID 29524189
- [Result] de Groot S, Enters-Weijnen CF, Geelhoed-Duijvestijn PH, Kanters TA. A cost of illness study of hypoglycaemic events in insulin-treated diabetes in the Netherlands. BMJ Open. 2018 Mar 25;8(3):e019864. doi: 10.1136/bmjopen-2017-019864. PMID 29581204
- [Result] Khunti K, Cigrovski Berkovic M, Ludvik B, Moberg E, Barner Lekdorf J, Gydesen H, Pedersen-Bjergaard U. Regional variations in definitions and rates of hypoglycaemia: findings from the global HAT observational study of 27 585 people with Type 1 and insulin-treated Type 2 diabetes mellitus. Diabet Med. 2018 May 5;35(9):1232-41. doi: 10.1111/dme.13662. Online ahead of print. PMID 29729048
- [Result] Pedersen-Bjergaard U, Alsifri S, Aronson R, Berkovic MC, Galstyan G, Gydesen H, Lekdorf JB, Ludvik B, Moberg E, Ramachandran A, Khunti K. Comparison of the HAT study, the largest global hypoglycaemia study to date, with similar large real-world studies. Diabetes Obes Metab. 2019 Apr;21(4):844-853. doi: 10.1111/dom.13588. Epub 2018 Dec 17. PMID 30456887
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com